CLINICAL TRIAL: NCT04071236
Title: A Phase I and Randomized Phase II Trial of Radium-223 Dichloride, M3814, &Amp; Avelumab in Advanced Metastatic Castrate-Resistant Prostate Cancer (mCRPC)
Brief Title: Radiation Medication (Radium-223 Dichloride) Versus Radium-223 Dichloride Plus Radiation Enhancing Medication (M3814) Versus Radium-223 Dichloride Plus M3814 Plus Avelumab (a Type of Immunotherapy) for Advanced Prostate Cancer Not Responsive to Hormonal Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-05620; NCI-2019-05620 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 202006062; 10301 (Other: Yale University Cancer Center LAO); 10301 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-Resistant Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Lymph Nodes; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Lymphatic Metastasis; Prostatic Neoplasms | interventions — avelumab; Specimen Handling; Magnetic Resonance Spectroscopy; peposertib; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (radium-223 dichloride) (Active Comparator): Patients receive radium-223 dichloride IV over 1 minute on day 1. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone scan, and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Radiation: Radium Ra 223 Dichloride
- Arm B (radium-223 dichloride, nedisertib) (Active Comparator): Patients receive radium-223 dichloride as in Arm A and peposertib PO or BID on days 3-26. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone scan, and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Peposertib; Other: Questionnaire Administration; Radiation: Radium Ra 223 Dichloride
- Arm C (radium-223 dichloride, nedisertib, avelumab) (Experimental): Patients receive radium-223 dichloride IV as in Arm A and peposertib PO QD or BID as in Arm B. Patients also receive avelumab IV over 60 minutes on days 1 and 15 of cycles 2-6. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone scan, and CT or MRI throughout the study.
  Interventions: Drug: Avelumab; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Peposertib; Other: Questionnaire Administration; Radiation: Radium Ra 223 Dichloride

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB 0010718C; MSB-0010718C; MSB0010718C
  Arms: Arm C (radium-223 dichloride, nedisertib, avelumab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib
  Arms: Arm B (radium-223 dichloride, nedisertib); Arm C (radium-223 dichloride, nedisertib, avelumab)
Other: Questionnaire Administration — Ancillary studies
Radiation: Radium Ra 223 Dichloride — Given IV
  Other Names: Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM RA-223 DICHLORIDE; Radium-223 Chloride; Radium-223 Dichloride; Xofigo

SUMMARY:
This phase I/II trial studies the best dose of M3814 when given together with radium-223 dichloride or with radium-223 dichloride and avelumab and to see how well they work in treating patients with castrate-resistant prostate cancer that had spread to other places in the body (metastatic). M3814 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radioactive drugs, such as radium-223 dichloride, may carry radiation directly to tumor cells and not harm normal cells. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. This study is being done to find out the better treatment between radium-223 dichloride alone, radium-223 dichloride in combination with M3814, or radium-223 dichloride in combination with both M3814 and avelumab, to lower the chance of prostate cancer growing or spreading in the bone, and if this approach is better or worse than the usual approach for advanced prostate cancer not responsive to hormonal therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of peposertib (M3814) in combination with radium-223 dichloride or in combination with radium-223 dichloride and avelumab in patients with advanced metastatic castrate-resistant prostate cancer (mCRPC) based on dose limiting toxicities (DLTs) in the doublet or triplet combinations. (Phase 1) II. Radiographic progression free survival (rPFS) will be evaluated based on both skeletal and extraskeletal progression following Prostate Cancer Working Group 3 (PCWG3) methodology. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine the time to the first symptomatic skeletal event [SSE]. II. To determine the safety of radium-223 dichloride, M3814, and avelumab combination treatment.

III. To observe and record anti-tumor activity. IV. To evaluate progression free survival (PFS) and overall survival (OS). V. To evaluate symptomatic skeletal events (SSE) per standardized case report form (CRF) distinguishing between pathologic and non-pathogenic fractures.

VI. To explore patient-reported symptomatic adverse events (AE) for tolerability of each treatment arm.

VII. To examine the radium-223 dichloride bio-distribution and absorbed dose in each bone metastatic lesions as well as elsewhere in the body including critical organs using dosimetry.

EXPLORATORY OBJECTIVES:

I. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES), and messenger ribonucleic acid (RNA) sequencing (RNAseq), in order to:

Ia. Identify potential predictive and prognostic biomarkers beyond any genomic alteration by which treatment may be assigned, and Ib. Identify resistance mechanisms using genomic deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

II. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

III. To bank plasma and peripheral immune cells from patients to assess predictive biomarkers of response at the Experimental Therapeutics Clinical Trials Network (ETCTN) biorepository at Nationwide Children's Hospital.

IV. To correlate change in level of total alkaline phosphatase, bone-specific alkaline phosphatase, and serum osteocalcin to rPFS and OS.

OUTLINE: This is a phase I, dose-escalation study of peposertib, followed by a phase II study. Patients are randomized to 1 of 3 arms.

ARM A: Patients receive radium-223 dichloride intravenously (IV) over 1 minute on day 1. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone scan, and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

ARM B: Patients receive radium-223 dichloride as in Arm A and peposertib orally (PO) once daily (QD) or twice daily (BID) on days 3-26. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone scan, and CT or MRI throughout the study.

ARM C: Patients receive radium-223 dichloride IV as in Arm A and peposertib PO QD or BID as in Arm B. Patients also receive avelumab IV over 60 minutes on days 1 and 15 of cycles 2-6. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone scan, and CT or MRI throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE 1: Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* PHASE 2: ECOG performance status =< 2 (Karnofsky >= 60%)
* Unless a patient has had orchiectomy by surgery, the patient is expected to be on antiandrogen therapy (ADT) for "medical castration". ADT needs to be maintained throughout the study. Testosterone level should be checked, and kept consistently lower than 50 ng/dL, similar to that obtained with bilateral orchiectomy
* Progressive castration-resistant prostate cancer with two or more skeletal metastases identified by 99mTC bone scintigraphy. One or more lymph node metastases allowed, but not mandatory. Lymph node metastases in each individually must measure less than 3 cm in the longest dimension. Visible visceral organ metastases are not allowed. A diagnosis of prostate cancer must have been histologically confirmed at any time point
* Baseline prostatic specific antigen (PSA) level of 1 ng/mL or higher with evidence of progressively increasing PSA values (two consecutive increases over the previous reference value)
* Progression after at least one of the following: abiraterone, enzalutamide, apalutamide, darolutamide, or taxane chemotherapy (docetaxel, cabazitaxel). There is no maximum number of prior therapies. Prior immunotherapies (for example, Sipuleucel-T or pembrolizumab) do not exclude the patient from participation
* Age >= 18 years. Castrate-resistant prostate cancer (CRPC) affects older adults and is rarely encountered in children and adolescents
* Life expectancy >= 6 months
* Albumin > 2.5 mg/dL
* Hemoglobin > 9 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (with the exception of < 3 mg/dL for patients with Gilbert's disease)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.5 x institutional ULN OR
* Glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy (with no medications prohibited by this protocol [e.g. drug-drug interactions]) with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy (with no medications prohibited by this protocol [e.g. drug-drug interactions]), if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load (with no medications prohibited by this protocol [e.g. drug-drug interactions])
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional classification. To be eligible for this trial, patients should be class 2B or better
* Concomitant use of physiologic corticosteroids is allowed
* Concomitant use of bisphosphonates is allowed (use of bone health agents is mandatory - either denosumab [preferred] or bisphosphonates)
* The effects of radium-223 dichloride, M3814, and avelumab on the developing human fetus are unknown. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of Radium-223 dichloride, M3814, and avelumab administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Patients must be able to swallow orally administered medication
* Patients with asymptomatic, treated brain metastases are permitted if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or CT scan) during the screening period

Exclusion Criteria:

* Active autoimmune conditions or patients on chronic immunosuppression due to underlying autoimmune condition
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients who have had previous hemibody external radiation
* Patients who have imminent/established spinal cord compression, pathological fracture in weight bearing bones or bone lesion with soft tissue component unless treated as appropriate with radiation and/or surgery before starting on trial
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to radium-223 dichloride, M3814, or avelumab
* Patients unable to discontinue medications or substances that are potent inhibitors, inducers or sensitive substrates of CYP3A4/5 or CYP2C19 prior to study treatment are ineligible.

  * Medications or substances that are strong inhibitors of CYP3A4/5 or CYP2C19 must be discontinued at least 1 week prior to first M3814 dose.
  * Medications or substances that are strong inducers of CYP3A4/5 or CYP2C19 must be stopped at least 3 weeks prior to the first M3814 dose.
  * Drugs mainly metabolized by CYP3A with a narrow therapeutic index (as judged by the Investigator or authorized designee) must be discontinued at least 1 day prior to first M3814 dose.
  * Note: Because the lists of these agents are constantly changing, it is important to regularly consult a frequently- updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the- counter medicine or herbal product.
* Radium-223 dichloride should not be given concurrently with abiraterone plus prednisone/prednisolone
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have an active infection requiring systemic treatment
* Patients must not use immunosuppressive medication =< 7 days of registration, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Patients who cannot discontinue concomitant H2 blockers or proton-pump inhibitors (PPIs). Patients may confer with the study doctor to determine if such medications can be discontinued. These must be discontinued >= 5 days prior to study treatment. Patients do not need to discontinue calcium carbonate
* Patients receiving sorivudine or any chemically related analogues (such as brivudine) are excluded
* Patients with a known history or present osteonecrosis of the jaw

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (Phase 1) | Up to 28 days
  Adverse events will be summarized as count and percentages, overall as well as by dose level/regimen, by severity, and by patient characteristics.
Radiographic progression free survival (rPFS) (Phase 2) | Date of randomization to date of scan showing either skeletal or extraskeletal progression following Prostate Cancer Clinical Trials Working Group 3 methodology or death, assessed up to 2 years
  Empirical survival probabilities will be estimated by the Kaplan-Meier (KM) product limit method by arms and the survival difference between arms will be compared by 1-sided log rank test.

SECONDARY OUTCOMES:
PFS | From date of randomization to the event of disease recurrence/progression or death due to any cause, assessed up to 2 years
  Will be similarly analyzed using the KM method, log rank test and univariate and multivariate Cox model as described for rPFS.
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 2 years
  OS will be similarly analyzed using the KM method, log rank test and univariate and multivariate Cox model as described for rPFS.
Symptomatic skeletal event (SSE) | Up to 2 years post treatment
  Wiil be assessed per standardized case report form distinguishing between pathologic and non-pathologic fractures. SSE rate will be estimated using the KM estimates with 95% confidence interval.
Incidence of toxicity and adverse events | Up to 2 years post treatment
  Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

OTHER OUTCOMES:
Quality of life | Up to 2 years post treatment
  The Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) data will be evaluated for data quality, to characterize baseline symptom status of patients on study and the change over time, to explore the development of symptomatic adverse events (AEs) and the change over time, and to explore the patient scores with clinician graded AEs. PRO-CTCAE data will be summarized descriptively as the number (percent) of patients reporting each grade for individual items. Comparisons between the two treatment arms will be performed on a per question basis.
Biomarker analysis | Up to 2 years post treatment
  Gleason score at baseline will be grouped as =< 6, 7 and >= 8. Prostate specific antigen (PSA) at baseline will be classified as =< 10, 10~20 and > 20 ng/mL. Categorical Gleason score, PSA will be summarized by counts and percentages. Fisher's exact test will be used to examine the distribution of Gleason score and PSA. Descriptive statistics will be used to summarize quantitative imaging/biomarker by arm. Multivariate Cox model will be applied to data across arms to examine the effect of Gleason score, pretreatment PSA, clinical stage etc. incorporated with adjusted hazard ratio reported with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Hiram A Gay, Principal Investigator — Yale University Cancer Center LAO
Locations (32):
- United States (32):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm